## Document 1 — Study Protocol (NAID-F)

**Cover Page** - Official Study Title: Risk of Anemia Development and Clinical Effects of Oral Iron Therapy in Women (18–55 Years) With Non-Anemic Iron Deficiency - NCT Number: [To be assigned] - Document Date: October 28, 2025

- **1. Study Identification** Organization's Unique Protocol ID: 2024-KAEK-22 Brief Title: Risk of Anemia and Effects of Oral Iron Therapy in Non-Anemic Iron-Deficient Women (18–55 Years) Acronym: NAID-F Study Type: Interventional Official Title: Risk of Anemia Development and Clinical Effects of Oral Iron Therapy in Women (18–55 Years) With Non-Anemic Iron Deficiency Secondary IDs: Other Identifier: E-14028348-302.14.02-985103 (Istanbul Univ.–Cerrahpasa Faculty of Medicine, Thesis Approval) Other Identifier: E-15916306-604.01-281470566 (Istanbul Provincial Health Directorate, Institutional Approval)
- **2. Study Status** Record Verification Date: October 2025 Overall Recruitment Status: Recruiting Study Start Date: September 01, 2025 (Actual) Primary Completion Date: January 01, 2026 (Anticipated) Study Completion Date: February 28, 2026 (Anticipated)
- **3. Sponsors and Collaborators** Responsible Party: Principal Investigator Investigator Name [Username]: Osman Demir, MD [odemir] Investigator Official Title: MD Investigator Affiliation: Istanbul University Cerrahpasa Name of Sponsor: Istanbul University Cerrahpasa Collaborators: Istanbul University Cerrahpasa
- **4. Oversight** U.S. FDA-Regulated Drug: No U.S. FDA-Regulated Device: No IND/IDE: No Human Subjects Protection Review: Approved Board Name: Istanbul University Cerrahpaşa Clinical Research Ethics Committee Approval Number: 2024-KAEK-22 Board Affiliation: Istanbul University Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Clinical Research Ethics Committee Board Contact: +90 (212) 414 32 52, kliniketik@iuc.edu.tr
- **5. Study Description** Brief Summary: This study investigates anemia risk and clinical effects of oral iron therapy in women aged 18–55 years with non-anemic iron deficiency. Conducted in two phases at Kağıthane 5 No'lu Family Health Center, Istanbul. Phase 1 (Observational Nutrition Intervention, 2 months): All participants receive dietary guidance to improve iron intake and absorption. Biweekly phone monitoring. Participants classified into five subgroups (ARM1-0 to ARM1-4) based on hematologic outcomes after 2 months. Phase 2 (Experimental Oral Iron Therapy, 1 month): Participants in ARM1-1 to ARM1-4 receive oral ferrous sulfate 80 mg/day. ARM1-0 participants maintain normal iron status and do not receive therapy.
- **6. Conditions** Non-Anemic Iron Deficiency Risk of Anemia Development Clinical Effects of Oral Iron Therapy Keywords: Iron Deficiency Without Anemia, Women 18–55 years, Hemoglobin, Ferritin, Symptom Scores, Prospective Cohort, Experimental Intervention, Iron Supplementation, Nutritional Intervention, Study Design
- **7. Study Design** Primary Purpose: Treatment Study Phase: N/A Interventional Study Model: Single Group Assignment Number of Arms: 1 Masking: None (Open Label) Allocation: Non-Randomized Enrollment: 60 (Anticipated) Arms and Interventions: Experimental: ARM 1 Nutritional Intervention with Post-Intervention Subgrouping (All participants receive 2-month dietary intervention; subgrouping based on lab outcomes; persistent iron deficiency participants receive 1-month oral elemental iron 80

- mg/day). Other: Dietary Intervention (2 months) iron-rich foods, absorption enhancement strategies, biweekly follow-up. Drug: Oral Elemental Iron (Ferrous Sulfate) 80 mg/day 1 month for persistent iron deficiency.
- **8. Outcome Measures Primary Outcome:** 1. Change from Baseline in Patient-Reported Iron Deficiency Symptom Scores (Baseline, Week 8, Week 12) **Secondary Outcomes:** 2. Hemoglobin and RBC indices (Baseline, Week 8, Week 12) 3. Serum Iron and TIBC (Baseline, Week 8, Week 12) 4. Incidence of progression to anemia after 2-month nutritional intervention (Week 8) 5. Hematologic response to 1-month oral iron therapy (Hb increase ≥1 g/dL; Week 8–12) 6. Ferritin response to 1-month oral iron therapy (Week 8–12) **Pre-specified Outcomes:** 7. Adherence to Nutritional Intervention (Week 0–8) 8. Adherence to Oral Iron Therapy (Week 8–12) 9. Incidence of Treatment-Related Adverse Events (Week 8–12)
- 9. Statistical Analysis Plan Data will be analyzed using repeated measures ANOVA for longitudinal comparisons of laboratory values and symptom scores. Participants will be stratified into five subgroups (ARM1-0 to ARM1-4) based on hematologic outcomes after 2 months. ANOVA comparisons will be performed across these five groups to assess differences in outcomes including hemoglobin, ferritin, RBC indices, serum iron, TIBC, and patient-reported symptom scores. Within-group changes over time will be analyzed using paired t-tests. Categorical data (proportions and percentages) will be analyzed using Chi-Square tests. Continuous variables will be summarized as mean  $\pm$  SD; categorical variables as counts and percentages. Subgroup analyses will focus on ARM1-1 to ARM1-4 participants who receive oral iron therapy. Sample size of 60 determined via G\*Power analysis ( $\alpha$ =0.05, 80% power). Missing data handled via multiple imputation if >5% missing.
- **10. Eligibility** Accepts Healthy Volunteers: No Sex: Female Age Limits: 18–55 years Inclusion Criteria: Female, 18–55 years, non-anemic iron deficiency (ferritin <15 μg/L), normal Hb, B12, folate, TSH, sT4, CRP <5 mg/L, informed consent. Exclusion Criteria: Pregnancy/postpartum, infection, malignancy, chronic disease, depression, chronic fatigue, kidney/heart disease, hematologic disorders, ongoing iron therapy.
- **11. Contacts and Locations** Central Contact Person: Osman Demir (+90 532 291 4470, osman.demir@iuc.edu.tr) Central Contact Backup: Ayşen Fenercioğlu (+90 537 964 5751, aysen.fenercioglu@iuc.edu.tr) Study Officials: Osman Demir (Principal Investigator), Kağıthane No.5 Family Health Center, Istanbul, Turkey; Ayşen Fenercioğlu (Study Director), Istanbul University Cerrahpaşa. Location: Kağıthane No.5 Family Health Center, Istanbul, Turkey (Recruiting)
- **12. IPD Sharing Statement** Plan to Share IPD: Undecided; to be determined post-study in accordance with ethics and participant privacy.
- **13. References and Additional Information** 1. World Health Organization. Guideline on the Use of Ferritin Concentrations to Assess Iron Status in Individuals and Populations. Geneva: WHO; 2020. 2. Soppi ET. Iron deficiency without anemia: a clinical challenge. Clin Case Rep. 2018;6:1082–1086. https://doi.org/10.1002/ccr3.1529 3. Balendran S, Forsyth C. Non-anaemic iron deficiency. Aust Prescr. 2021;44(6):193–196. doi:10.18773/austprescr.2021.052 4. World Health Organization & FAO. Guidelines on Food Fortification with Micronutrients. Geneva: WHO Press; 2006. 5. Skolmowska D, Glabska D, Kolota A, Guzek D. Effectiveness of dietary interventions to treat iron-deficiency anemia in women: a systematic review. Nutrients. 2022;14:2724. https://doi.org/10.3390/nu14132724 6. Clenin G. Treatment of iron deficiency without anaemia. Swiss Med Wkly. 2017;147:w14434. 7. British Society for Haematology. Guideline for the Laboratory Diagnosis of Iron Deficiency in Adults and Children. Br J Haematol. 2022;196:523–529. 8. Houston BL, Hurrie D, Graham J, et al. Efficacy of iron supplementation

on fatigue in non-anemic iron-deficient adults: systematic review. BMJ Open. 2018;8:e019240. 9. Miles LF, Litton E, Imberger G, Story D. Intravenous iron therapy for non-anaemic, iron-deficient adults. Cochrane Database Syst Rev. 2019;12:CD013084. 10. da Silva Lopes K, Yamaji N, Rahman MO, et al. Nutrition-specific interventions for preventing and controlling anaemia: overview of systematic reviews. Cochrane Database Syst Rev. 2021;9:CD013092.